CLINICAL TRIAL: NCT00573274
Title: Pilot Study Measuring Cardiac Output and Stroke Volume Using Non-Invasive Thoracic Impedance With the Physioflow Impedance Device in Pregnant Patients Undergoing Cesarean Section Under Spinal Anesthesia
Brief Title: Measuring Cardiac Output and Stroke Volume Using the Physioflow Impedance Device in Pregnant Patients
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Eric Kong You-Ten, Mount Sinai Hospital
Other Study IDs: 07-09; 07-0225-E
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Hypotension
Keywords: Cesarean section; Cardiac Output; Physioflow; Cardiography, Impedance
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Elective cesarean section patients
  Interventions: Device: Physioflow Impedance

INTERVENTIONS:
Device: Physioflow Impedance — 6 ECG leads applied to the neck and thorax for the duration of surgery (approximately 1 hour).

SUMMARY:
Pregnant patients having a cesarean section (CS) under spinal anesthesia experience a variety of hemodynamic changes, such as hypotension due to decreases in cardiac output (CO), stroke volume (SV) and/or systemic vascular resistance (SVR). Measurement of these hemodynamic parameters classically requires insertion of a pulmonary artery catheter (PAC) into the heart. However, this invasive method carries significant complications and its use is now reserved for the more critically ill patients. We hypothesize that the Physioflow Impedance device can be used as a reliable non-invasive monitor to measure hemodynamic parameters during elective CS under spinal anesthesia.

DETAILED DESCRIPTION:
The Physioflow Impedance device employs a continuous non-invasive method of measuring ten cardiac hemodynamic parameters including flow, resistance, contractility and fluid content. It involves the application of electrocardiogram (ECG) leads on the neck and the thorax to measure resistance of pulsatile blood flow. Its benefits are that it is non-invasive, low cost, and easy to operate. Thoracic impedance has been validated against the gold standard method of PAC. Although the Physioflow device has been validated in non-pregnant patients, its use in pregnant patients is very limited.

Moderate to severe hypotension, experienced by these awake patients, can cause significant undesirable symptoms of dizziness, shortness of breath, nausea and vomiting, and also compromise fetal well-being. The etiology of hypotension is multi-factorial,and it is postulated that decreases in cardiac output (CO), stroke volume (SV) and/or systemic vascular resistance (SVR) may precede decreases in blood pressure. Continuous measurement of CO and SV by the Physioflow Impedance device may provide a better understanding of the cause of hypotension so that future management of these patients may include pharmacological interventions used prior to hypotension in order to avoid any undesirable symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective cesarean section
* Women classified as ASA 1 & 2

Exclusion Criteria:

* Patients unable to communicate in English
* Patients with significant cardiac disease
* Height less than 4 feet or greater than 7 feet
* Weight less than 67 lbs or greater than 341 lbs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers having an elective cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Continuous measurement of cardiac output (CO), stroke volume (SV) and/or systemic vascular resistance (SVR) changes. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kong Eric You-Ten, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada